CLINICAL TRIAL: NCT05608031
Title: Which Value of 6th Month EWL% After Sleeve Gastrectomy is Needed to Get a Better Sleep Quality?
Brief Title: 6th Month EWL% After Sleeve Gastrectomy to Get a Better Sleep Quality
Status: Completed | Type: Observational
Sponsor: Umraniye Education and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Fatih Basak, Clinical Associate Professor, Umraniye Education and Research Hospital
Other Study IDs: Obesity-Sleep-Quality
Record Dates: First submitted 2022-11-01; First posted 2022-11-07 (Actual); Last update posted 2022-11-07 (Actual); Status verified 2022-11

CONDITIONS: Sleep Disturbance; Obesity, Severe; Surgery
Keywords: Laparoscopic sleeve gastrectomy; Pittsburgh sleep quality index; Obesity
MeSH Terms: conditions — Parasomnias; Obesity, Morbid; Obesity | interventions — Weights and Measures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- bariatric surgery: A cross-sectional study was conducted among patients that underwent bariatric surgery (laparoscopic sleeve gastrectomy). Sleep quality was assessed using the Pittsburgh sleep quality index (PSQI) scale preoperatively and at the 6th postoperative month.
  Interventions: Other: Pittsburgh sleep quality index (PSQI) scale

INTERVENTIONS:
Other: Pittsburgh sleep quality index (PSQI) scale — Pittsburgh Sleep Quality Index (PSQI) (6), a self-report questionnaire comprising seven component scores (subjective sleep quality, sleep latency, duration of sleep, sleep efficiency habits, sleep disturbances, use of sleeping medication, and daytime dysfunction), was used to evaluate sleep quality over the last month.

SUMMARY:
Obesity, caused by caloric intake over output, has become a global health problem. The relationship between sleep and obesity is widely discussed in the literature. Little is known regarding the compliance of sleep quality and patients' weight loss. This study aimed to review how sleep quality is affected by bariatric surgery, examine whether compliance with sleep quality can be predicted after bariatric surgery, and assess its correlation with excess weight loss.

DETAILED DESCRIPTION:
A cross-sectional study was conducted among patients that underwent bariatric surgery (laparoscopic sleeve gastrectomy). Sleep quality was assessed using the Pittsburgh sleep quality index (PSQI) scale preoperatively and at the 6th postoperative month. Survey data were recorded and PSQI scores were calculated. A PSQI global score above 5 indicates poor sleep quality. The participants were divided into two groups good sleep quality and poor sleep quality. Descriptive statistics and Spearman correlations were applied. Logistic regression analysis was performed to predict sleep quality.

ELIGIBILITY:
Inclusion Criteria:

Patients who underwent LSG for morbid obesity after being considered suitable for bariatric surgery by multidisciplinary evaluation were included in this study. Patients with aged 18-65 years, BMI > 40 and BMI > 35 and comorbid disease were included.

Exclusion Criteria:

Patients treated for sleep disorders have been excluded.

Age Groups: Child, Adult, Older Adult
Study Population: Demographic parameters of the patients, preoperative and follow-up weight, body mass index (BMI), percentage of excess weight loss (EWL%), and percentage of excess BMI loss (EBMI%) were noted. The Pittsburgh Sleep Quality Index (PSQI) questionnaire was applied to all patients preoperatively. Survey data were recorded and PSQI scores were calculated. Appropriate nutrition and physical activity programs were administered to all patients postoperatively under the control of a nutritionist.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
good sleep quality | 6 months
  A PSQI global score above 5 indicates poor sleep quality.
poor sleep quality | 6 months
  A PSQI global score above 5 indicates poor sleep quality.

CONTACTS AND LOCATIONS:
Locations (1):
- Umraniye Education and Research Hospital, Istanbul, Ümraniye, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No